CLINICAL TRIAL: NCT04640168
Title: A Multicenter, Adaptive, Randomized Blinded Controlled Trial of the Safety and Efficacy of Investigational Therapeutics for the Treatment of COVID-19 in Hospitalized Adults (ACTT-4)
Brief Title: Adaptive COVID-19 Treatment Trial 4 (ACTT-4)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20-0006 ACTT-4
Record Dates: First submitted 2020-11-19; First posted 2020-11-23 (Actual); Results first posted 2022-06-28 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2021-04

CONDITIONS: COVID-19
Keywords: ACTT; Adaptive; COVID-19; Efficacy; Multicenter; novel coronavirus; Safety
MeSH Terms: conditions — COVID-19 | interventions — baricitinib; Dexamethasone; remdesivir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Remdesivir plus Baricitinib (Experimental): 200 mg of remdesivir administered intravenously on Day 1, followed by a 100 mg once-daily maintenance dose of remdesivir while hospitalized for up to a 10-day total course; 4 mg of baricitinib administered as 2 tablets taken orally daily while hospitalized for up to a 14-day total course; and dexamethasone placebo administered as an intravenous injection daily while hospitalized for up to a 10-day total course.
  Interventions: Drug: Baricitinib; Other: Placebo; Drug: Remdesivir
- Remdesivir plus Dexamethasone (Experimental): 200 mg of remdesivir administered intravenously on Day 1, followed by a 100 mg once-daily maintenance dose of remdesivir while hospitalized for up to a 10-day total course; baricitinib placebo administered as 2 tablets taken orally daily while hospitalized for up to a 14-day total course; and 6 mg of dexamethasone administered as an intravenous injection daily while hospitalized for up to a 10-day total course.
  Interventions: Drug: Dexamethasone; Other: Placebo; Drug: Remdesivir

INTERVENTIONS:
Drug: Baricitinib — Baricitinib is a Janus kinase (JAK) inhibitor with the chemical name [1-(ethylsulfonyl)-3-(4-(7Hpyrrolo(2,3-d)pyrimidin-4-yl)-1H-pyrazol-1-yl)azetidin-3-yl]acetonitrile. Each tablet contains 2 mg of baricitinib and the following inactive ingredients: croscarmellose sodium, magnesium stearate, mannitol, microcrystalline cellulose, ferric oxide, lecithin (soya), polyethylene glycol, polyvinyl alcohol, talc and titanium dioxide.
  Arms: Remdesivir plus Baricitinib
Drug: Dexamethasone — Dexamethasone Sodium Phosphate Injection, USP, is an adrenocortical steroid anti-inflammatory drug. It is a water-soluble inorganic ester of dexamethasone. Each mL contains dexamethasone sodium phosphate equivalent to dexamethasone phosphate 4 mg or dexamethasone 3.33 mg; benzyl alcohol 10 mg added as preservative; sodium citrate dihydrate 11 mg; sodium sulfite 1 mg as an antioxidant.
  Arms: Remdesivir plus Dexamethasone
Other: Placebo — Placebo matching oral baricitinib or intravenous dexamethasone.
Drug: Remdesivir — Drug remdesivir is a single diastereomer monophosphoramidate prodrug designed for the intracellular delivery of a modified adenine nucleoside analog GS-441524. In addition to the active ingredient, the lyophilized formulation of remdesivir contains the following inactive ingredients: water for injection, sulfobutylether beta-cyclodextrin sodium (SBECD), and hydrochloric acid and/or sodium hydroxide.

SUMMARY:
ACTT-4 will evaluate the combination of baricitinib and remdesivir compared to dexamethasone and remdesivir. Subjects will be assessed daily while hospitalized. If the subjects are discharged from the hospital, they will have a study visit at Days 15, 22, and 29. For discharged subjects, it is preferred that the Day 15 and 29 visits are in person to obtain safety laboratory tests, oropharyngeal (OP) swabs, plasma (Day 29), and serum for secondary research as well as clinical outcome data. However, if infection control or other restrictions limit the ability of the subject to return to the clinic, these visits may be conducted by phone, and only clinical data will be obtained. The Day 22 visit does not have laboratory tests or collection of samples and is conducted by phone. The primary objective is to evaluate the clinical efficacy of baricitinib + remdesivir versus dexamethasone + remdesivir as assessed by the mechanical ventilation free survival by Day 29.

DETAILED DESCRIPTION:
This study is an adaptive randomized double-blind placebo-controlled trial to evaluate the safety and efficacy of novel therapeutic agents in hospitalized adults diagnosed with COVID-19. The study is a multicenter trial that will be conducted in up to approximately 100 sites globally. The study will compare different investigational therapeutic agents to a control arm. New arms can be introduced according to scientific and public health needs. There will be interim monitoring to allow early stopping for futility, efficacy, or safety. If one therapy proves to be efficacious, then this treatment may become the control arm for comparison(s) with new experimental treatment(s). Any such change would be accompanied by an updated sample size. This adaptive platform is used to rapidly evaluate different therapeutics in a population of those hospitalized with moderate to severe COVID-19. The platform will provide a common framework sharing a similar population, design, endpoints, and safety oversight. New stages with new therapeutics can be introduced. One independent Data and Safety Monitoring Board (DSMB) will actively monitor interim data in all stages to make recommendations about early study closure or changes to study arms.

ACTT-4 will evaluate the combination of baricitinib and remdesivir compared to dexamethasone and remdesivir. Subjects will be assessed daily while hospitalized. If the subjects are discharged from the hospital, they will have a study visit at Days 15, 22, and 29. For discharged subjects, it is preferred that the Day 15 and 29 visits are in person to obtain safety laboratory tests, oropharyngeal (OP) swabs, plasma (Day 29), and serum for secondary research as well as clinical outcome data. However, if infection control or other restrictions limit the ability of the subject to return to the clinic, these visits may be conducted by phone, and only clinical data will be obtained. The Day 22 visit does not have laboratory tests or collection of samples and is conducted by phone.

All subjects will undergo a series of efficacy, safety, and laboratory assessments. Safety laboratory tests and blood (serum and plasma) research samples and oropharyngeal (OP) swabs will be obtained on Days 1 (prior to infusion) and Days 3, 5, 8, and 11 (while hospitalized). OP swabs and blood (serum only) plus safety laboratory tests will be collected on Day 15 and 29 (if the subject attends an in-person visit or are still hospitalized).

The primary objective is to evaluate the clinical efficacy of baricitinib + remdesivir versus dexamethasone + remdesivir as assessed by the mechanical ventilation free survival by Day 29. The key secondary objective is to evaluate the clinical efficacy of baricitinib + remdesivir versus dexamethasone + remdesivir according to clinical status (8-point ordinal scale) at Day 15.

Contacts:

20-0006 Central Contact

Telephone: 1 (301) 7617948

Email: DMIDClinicalTrials@niaid.nih.gov

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized with symptoms suggestive of COVID-19.
2. Subject (or legally authorized representative) provides informed consent prior to initiation of any study procedures and understands and agrees to comply with planned study procedures.
3. Male or non-pregnant female adult > / = 18 years of age at time of enrollment.
4. Illness of any duration and has laboratory-confirmed SARS-CoV-2 infection as determined by polymerase chain reaction (PCR) or other commercial or public health assay (e.g. NAAT, antigen test) in any respiratory specimen or saliva < / = 14 days prior to randomization.
5. Within the 7 days prior to randomization requiring new use of supplemental oxygen (or increased oxygen requirement if on chronic oxygen) and requires at the time of randomization low or high flow oxygen devices or use of non-invasive mechanical ventilation (ordinal scale category 5 or 6).
6. Women of childbearing potential must agree to either abstinence or use at least one primary form of contraception not including hormonal contraception from the time of screening through Day 29.
7. Agrees not to participate in another blinded clinical trial (both pharmacologic and other types of interventions) for the treatment of COVID-19 through Day 29.

Exclusion Criteria:

1. Prior enrollment in ACTT-3 or ACTT-4. Note: this includes subjects whose participation in ACTT was terminated early.
2. On invasive mechanical ventilation at the time of randomization (ordinal scale category 7).
3. Anticipated discharge from the hospital or transfer to another hospital which is not a study site within 72 hours of randomization.
4. Positive test for influenza virus during the current illness (influenza testing is not required by protocol).
5. Subjects with a low glomerular filtration rate (eGFR), specifically:

   1. Subjects with an eGFR 15-30 mL/min are excluded unless in the opinion of the PI, the potential benefit of participation outweighs the potential risk of study participation.
   2. All subjects with an eGFR <15 mL/min
   3. All subjects on hemodialysis and/or hemofiltration at screening, irrespective of eGFR are excluded.
6. Neutropenia (absolute neutrophil count <700 cells/microliter, 0.7 x 10^3/microliter).
7. Lymphopenia (absolute lymphocyte count <200 cells/microliter, 0.20 x 10^3/microliter).
8. Received five or more doses of remdesivir including the loading dose, outside of the study as treatment for COVID-19.
9. Pregnancy or breast feeding (lactating women who agree to discard breast milk from Day 1 until two weeks after the last study product is given are not excluded).
10. Allergy to any study medication.
11. Received convalescent plasma or intravenous immunoglobulin [IVIg] for COVID-19, the current illness for which they are being enrolled.
12. Received any of the following in the two weeks prior to screening as treatment of COVID-19:

    * More than one dose of baricitinib for the treatment of COVID-19;
    * Other small molecule tyrosine kinase inhibitors (e.g. imatinib, gefitinib, acalabrutinib, etc.);
    * monoclonal antibodies targeting cytokines (e.g., TNF inhibitors, anti-interleukin-1 [IL-1], anti-IL-6 [tocilizumab or sarilumab], etc.);
    * monoclonal antibodies targeting T-cells or B-cells as treatment for COVID-19. Note: receipt of anti-SARS-CoV-2 monoclonal antibody (mAb) prior to enrollment (e.g. bamlanivimab) for their current COVID-19 illness is not exclusionary
13. Use of probenecid that cannot be discontinued at study enrollment.
14. Received 6 mg or more of dexamethasone by mouth (po) or Intravenous (IV) (or equivalent for other glucocorticoids) in one day, on more than one day, in the 7 days prior to time of randomization. Note: 6 mg dexamethasone dose equivalents include 40 mg prednisone, 32 mg methylprednisolone and 160 mg hydrocortisone.
15. Received > / = 20 mg/day of prednisone po or IV (or equivalent for other glucocorticoids) for > / = 14 consecutive days in the 4 weeks prior to screening.
16. Have diagnosis of current active or latent tuberculosis (TB), if known, treated for less than 4 weeks with appropriate therapy (by history only, no screening required).
17. Serious infection (besides COVID-19), immunosuppressive state, or immunosuppressive medications that in the opinion of the investigator could constitute a risk when taking baricitinib or dexamethasone.
18. Have received any live vaccine (that is, live attenuated) within 4 weeks before screening, or intend to receive a live vaccine (or live attenuated) during the study. Note: Use of non-live (inactivated) vaccinations including SARS-CoV-2 vaccine is allowed for all subjects.
19. Had a known Venous thromboembolism (VTE)(deep vein thrombosis [DVT] or pulmonary embolism [PE]) during the current COVID-19 illness.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1010 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2021-05-18 (Actual); Study Completion 2021-06-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (72):
- United States (61):
  - University of Alabama at Birmingham School of Medicine - Infectious Disease, Birmingham, Alabama
  - UCSF Fresno Center for Medical Education and Research - Clinical Research Center, Fresno, California
  - University of California San Diego Health - Jacobs Medical Center, La Jolla, California
  - University of California Los Angeles Medical Center - Westwood Clinic, Los Angeles, California
  - University of California Irvine Medical Center - Infectious Disease, Orange, California
  - VA Palo Alto Health Care System - Infectious Diseases, Palo Alto, California
  - University of California Davis Medical Center - Internal Medicine - Infectious Disease, Sacramento, California
  - Kaiser Permanente San Diego Medical Center, San Diego, California
  - Naval Medical Center San Diego - Infectious Disease Clinic, San Diego, California
  - University of California San Francisco - Zuckerberg San Francisco General Hospital - Division of Human Immunodeficiency Virus, Infectious Disease, and Global Medicine, San Francisco, California
  - Stanford University - Stanford Hospital and Clinics - Pediatrics - Infectious Diseases, Stanford, California
  - Cedars Sinai Medical Center, West Hollywood, California
  - VA Eastern Colorado Health Care System, Aurora, Colorado
  - Denver Health Division of Hospital Medicine - Main Campus, Denver, Colorado
  - Georgetown University Medical Center - Division of Infectious Diseases, Washington D.C., District of Columbia
  - University of Florida Health - Shands Hospital - Division of Infectious Diseases and Global Medicine, Gainesville, Florida
  - University of Florida Health - Jacksonville - Department of Emergency Medicine, Jacksonville, Florida
  - University of Miami Miller School of Medicine - Infectious Diseases, Miami, Florida
  - Emory Vaccine Center - The Hope Clinic, Decatur, Georgia
  - Atlanta VA Medical Center - Infectious Diseases Clinic, Decatur, Georgia
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Northwestern Hospital - Infectious Disease, Chicago, Illinois
  - University of Illinois at Chicago College of Medicine - Division of Infectious Diseases, Chicago, Illinois
  - University of Iowa Hospitals & Clinics - Department of Internal Medicine, Iowa City, Iowa
  - Tulane University - Section of Pulmonary Diseases, Critical Care, and Environmental Medicine, New Orleans, Louisiana
  - University of Maryland School of Medicine - Center for Vaccine Development - Baltimore, Baltimore, Maryland
  - Johns Hopkins Hospital - Medicine - Infectious Diseases, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - National Institutes of Health - Clinical Center, National Institute of Allergy and Infectious Diseases Laboratory Of Immunoregulation, Clinical Research Section, Bethesda, Maryland
  - Massachusetts General Hospital - Infectious Diseases, Boston, Massachusetts
  - University of Massachusetts Medical School - Infectious Diseases and Immunology, Worcester, Massachusetts
  - University of Michigan - Infectious Disease Clinic at Taubman Center, Ann Arbor, Michigan
  - University of Minnesota Medical Center, Fairview - Infectious Diseases and International Medicine, Minneapolis, Minnesota
  - Saint Louis University - Center for Vaccine Development, St Louis, Missouri
  - University of Nebraska Medical Center - Infectious Diseases, Omaha, Nebraska
  - CHI Health Creighton University Medical Center - Bergan Mercy - Pulmonary Medicine, Omaha, Nebraska
  - Atlantic Health System - Morristown Medical Center, Morristown, New Jersey
  - University of New Mexico Clinical and Translational Science Center, Albuquerque, New Mexico
  - New York University School of Medicine - Langone Medical Center - Microbiology - Parasitology, New York, New York
  - University of Rochester Medical Center - Vaccine Research Unit, Rochester, New York
  - Montefiore Medical Center - Infectious Diseases, The Bronx, New York
  - Duke Human Vaccine Institute - Duke Vaccine and Trials Unit, Durham, North Carolina
  - Womack Army Medical Center - Pulmonary and Respiratory Services, Fort Bragg, North Carolina
  - University of Oklahoma Health Science Center - Surgery, Oklahoma City, Oklahoma
  - Kaiser Permanente Northwest - Center for Health Research, Portland, Oregon
  - Penn State Health Milton S. Hershey Medical Center - Division of Infectious Diseases, Hershey, Pennsylvania
  - Hospital of the University of Pennsylvania - Infectious Diseases, Philadelphia, Pennsylvania
  - University of Pittsburgh - Medicine - Infectious Diseases, Pittsburgh, Pennsylvania
  - Baylor Scott & White Health - Baylor University Medical Center - North Texas Infectious Disease Consultants, Dallas, Texas
  - University of Texas Southwestern Medical Center - Internal Medicine - Infectious Diseases, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch - Division of Infectious Disease, Galveston, Texas
  - Methodist Hospital - Houston, Houston, Texas
  - Baylor College of Medicine - Molecular Virology and Microbiology, Houston, Texas
  - University of Texas Health Science Center at San Antonio - Infectious Diseases, San Antonio, Texas
  - University of Utah - Infectious Diseases, Salt Lake City, Utah
  - University of Virginia - Acute Care Surgery, Charlottesville, Virginia
  - Naval Medical Center Portsmouth - Infectious Disease Division, Portsmouth, Virginia
  - EvergreenHealth Infectious Disease Service, Kirkland, Washington
  - Providence Sacred Heart Medical Center, Spokane, Washington
  - Madigan Army Medical Center - Infectious Disease Clinic, Tacoma, Washington
- Japan (2):
  - Tokyo Medical and Dental University - Medical Hospital - Department of Respiratory Medicine, Tokyo
  - National Center for Global Health and Medicine Hospital - Disease Control and Prevention Center, Tokyo
- Mexico (2):
  - Instituto Nacional de Ciencias Medicas y Nutrición Salvador Zubirán - Departamento de Infectologia, Mexico City
  - Instituto Nacional de Enfermedades Respiratorias (INER) - Ismael Cosío Villegas, Mexico City
- Singapore (5):
  - National University Health System - Division of Infectious Diseases, Singapore
  - National University Health System - Alexandra Hospital - Division of Infectious Diseases, Singapore
  - National Centre for Infectious Diseases, Singapore
  - Changi General Hospital - Clinical Trials and Research Unit (CTRU), Singapore
  - Ng Teng Fong General Hospital - Infectious Disease Service, Singapore
- South Korea (2):
  - Seoul National University Bundang Hospital - Division of Infectious Diseases, Bundang-gu Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul, Jongno-gu

REFERENCES:
- [Derived] Potter GE, Bonnett T, Rubenstein K, Lindholm DA, Rapaka RR, Doernberg SB, Lye DC, Mularski RA, Hynes NA, Kline S, Paules CI, Wolfe CR, Frank MG, Rouphael NG, Deye GA, Sweeney DA, Colombo RE, Davey RT Jr, Mehta AK, Whitaker JA, Castro JG, Amin AN, Colombo CJ, Levine CB, Jain MK, Maves RC, Marconi VC, Grossberg R, Hozayen S, Burgess TH, Atmar RL, Ganesan A, Gomez CA, Benson CA, Lopez de Castilla D, Ahuja N, George SL, Nayak SU, Cohen SH, Lalani T, Short WR, Erdmann N, Tomashek KM, Tebas P. Temporal Improvements in COVID-19 Outcomes for Hospitalized Adults: A Post Hoc Observational Study of Remdesivir Group Participants in the Adaptive COVID-19 Treatment Trial. Ann Intern Med. 2022 Dec;175(12):1716-1727. doi: 10.7326/M22-2116. Epub 2022 Nov 29. PMID 36442063
- [Derived] Wolfe CR, Tomashek KM, Patterson TF, Gomez CA, Marconi VC, Jain MK, Yang OO, Paules CI, Palacios GMR, Grossberg R, Harkins MS, Mularski RA, Erdmann N, Sandkovsky U, Almasri E, Pineda JR, Dretler AW, de Castilla DL, Branche AR, Park PK, Mehta AK, Short WR, McLellan SLF, Kline S, Iovine NM, El Sahly HM, Doernberg SB, Oh MD, Huprikar N, Hohmann E, Kelley CF, Holodniy M, Kim ES, Sweeney DA, Finberg RW, Grimes KA, Maves RC, Ko ER, Engemann JJ, Taylor BS, Ponce PO, Larson L, Melendez DP, Seibert AM, Rouphael NG, Strebe J, Clark JL, Julian KG, de Leon AP, Cardoso A, de Bono S, Atmar RL, Ganesan A, Ferreira JL, Green M, Makowski M, Bonnett T, Beresnev T, Ghazaryan V, Dempsey W, Nayak SU, Dodd LE, Beigel JH, Kalil AC; ACTT-4 Study Group. Baricitinib versus dexamethasone for adults hospitalised with COVID-19 (ACTT-4): a randomised, double-blind, double placebo-controlled trial. Lancet Respir Med. 2022 Sep;10(9):888-899. doi: 10.1016/S2213-2600(22)00088-1. Epub 2022 May 23. PMID 35617986
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the participating sites from those admitted with symptoms of COVID-19 confirmed by PCR. Enrollment occurred between December 2, 2020 and April 13, 2021.
Groups:
- Remdesivir Plus Baricitinib: 200 mg of remdesivir administered intravenously on Day 1, followed by a 100 mg once-daily maintenance dose of remdesivir while hospitalized for up to a 10-day total course; 4 mg of baricitinib administered as 2 tablets taken orally daily while hospitalized for up to a 14-day total course; and dexamethasone placebo administered as an intravenous injection daily while hospitalized for up to a 10-day total course.
  Baricitinib: Baricitinib is a Janus kinase (JAK) inhibitor with the chemical name [1-(ethylsulfonyl)-3-(4-(7Hpyrrolo(2,3-d)pyrimidin-4-yl)-1H-pyrazol-1-yl)azetidin-3-yl]acetonitrile. Each tablet contains 2 mg of baricitinib and the following inactive ingredients: croscarmellose sodium, magnesium stearate, mannitol, microcrystalline cellulose, ferric oxide, lecithin (soya), polyethylene glycol, polyvinyl alcohol, talc and titanium dioxide.
  Placebo: Placebo matching intravenous dexamethasone.
  Remdesivir: Drug remdesivir is a single diastereomer monophosphoramidate prodrug designed for the intracellular delivery of a modified adenine nucleoside analog GS-441524. In addition to the active ingredient, the lyophilized formulation of remdesivir contains the following inactive ingredients: water for injection, sulfobutylether beta-cyclodextrin sodium (SBECD), and hydrochloric acid and/or sodium hydroxide.
- Remdesivir Plus Dexamethasone: 200 mg of remdesivir administered intravenously on Day 1, followed by a 100 mg once-daily maintenance dose of remdesivir while hospitalized for up to a 10-day total course; baricitinib placebo administered as 2 tablets taken orally daily while hospitalized for up to a 14-day total course; and 6 mg of dexamethasone administered as an intravenous injection daily while hospitalized for up to a 10-day total course.
  Dexamethasone: Dexamethasone Sodium Phosphate Injection, USP, is an adrenocortical steroid anti-inflammatory drug. It is a water-soluble inorganic ester of dexamethasone. Each mL contains dexamethasone sodium phosphate equivalent to dexamethasone phosphate 4 mg or dexamethasone 3.33 mg; benzyl alcohol 10 mg added as preservative; sodium citrate dihydrate 11 mg; sodium sulfite 1 mg as an antioxidant.
  Placebo: Placebo matching oral baricitinib.
  Remdesivir: Drug remdesivir is a single diastereomer monophosphoramidate prodrug designed for the intracellular delivery of a modified adenine nucleoside analog GS-441524. In addition to the active ingredient, the lyophilized formulation of remdesivir contains the following inactive ingredients: water for injection, sulfobutylether beta-cyclodextrin sodium (SBECD), and hydrochloric acid and/or sodium hydroxide.
Period: Overall Study
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Dexamethasone
Started | 516 | 494
Treated | 503 | 482
ITT and Modified ITT Population | 516 | 494
As Treated Population | 503 | 482
Completed | 495 | 475
Not Completed | 21 | 19
Not completed — Withdrawal by Subject | 8 | 7
Not completed — Lost to Follow-up | 1 | 0
Not completed — Enrolled but not treated | 12 | 12

BASELINE CHARACTERISTICS:
Population: The population includes all participants enrolled.
Groups:
- Total: Total of all reporting groups
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Dexamethasone | Total
Number analyzed (Participants) | 516 | 494 | 1010
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 345 | 330 | 675
  >=65 years | 171 | 164 | 335
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.2 (14.3) | 58.5 (13.7) | 58.3 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 216 | 204 | 420
  Male | 300 | 290 | 590
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 188 | 159 | 347
  Not Hispanic or Latino | 318 | 318 | 636
  Unknown or Not Reported | 10 | 17 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 8 | 10 | 18
  Asian | 35 | 35 | 70
  Native Hawaiian or Other Pacific Islander | 1 | 4 | 5
  Black or African American | 94 | 94 | 188
  White | 307 | 281 | 588
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 68 | 68 | 136
Region of Enrollment [Number; unit: participants]
  South Korea | 13 | 11 | 24
  Singapore | 2 | 2 | 4
  United States | 474 | 453 | 927
  Japan | 0 | 3 | 3
  Mexico | 27 | 25 | 52

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Participants Not Meeting Criteria for One of the Following Two Ordinal Scale Categories at Any Time: 8) Death; 7) Hospitalized, on Invasive Mechanical Ventilation or Extracorporeal Membrane Oxygenation (ECMO)
Description: Mechanical ventilation-free survival was assessed through Day 29, defined as the proportion of participants who had not died nor were hospitalized on invasive mechanical ventilation or ECMO as of Day 29. Results are reported as Kaplan Meier estimates.
Time Frame: Day 1 through Day 29
Population: The modified intention-to-treat (mITT) population includes all participants who were randomized. mITT participants were classified by their randomized treatment assignment and their baseline ordinal score, which is not necessarily equivalent to the disease severity stratum to which the participant was randomized at enrollment. One participant was excluded from mITT analyses due to a baseline ordinal score of 4.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Dexamethasone
Number analyzed (Participants) | 515 | 494
Proportion of participants | 0.87 [0.84 to 0.90] | 0.88 [0.84 to 0.90]
Statistical Analysis 1: Comparison: Remdesivir Plus Baricitinib vs Remdesivir Plus Dexamethasone; Test type: Superiority; p = 0.909, Chi-squared

2. Secondary Outcome: Change From Baseline in Alanine Aminotransferase (ALT)
Description: Blood to evaluate ALT was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge.
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: The safety population includes all treated participants with available data at baseline and the post baseline assessment point, analyzed as treated.
Measure: Mean (95% Confidence Interval); unit: Units/Liter (U/L)
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Dexamethasone
Number analyzed (Participants) | 483 | 458
Units/Liter (U/L)
  Day 3 | 1.1 [-0.9 to 3.1] | 4.3 [1.2 to 7.4]
  Day 5: number analyzed (Participants) | 366 | 342
  Day 5 | 6.0 [0.8 to 11.2] | 15.9 [11.6 to 20.1]
  Day 8: number analyzed (Participants) | 205 | 193
  Day 8 | 4.7 [-5.9 to 15.3] | 16.1 [2.6 to 29.7]
  Day 11: number analyzed (Participants) | 127 | 115
  Day 11 | 5.6 [-2.0 to 13.2] | 15.5 [4.1 to 26.9]
  Day 15: number analyzed (Participants) | 203 | 183
  Day 15 | 7.1 [-1.1 to 15.2] | 8.2 [-3.3 to 19.8]
  Day 29: number analyzed (Participants) | 220 | 191
  Day 29 | -3.8 [-16.3 to 1.0] | 1.1 [-26.3 to 18.5]

3. Secondary Outcome: Change From Baseline in Aspartate Aminotransferase (AST)
Description: Blood to evaluate AST was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge.
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: U/L
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Dexamethasone
Number analyzed (Participants) | 482 | 458
U/L
  Day 3 | -5.9 [-8.1 to -3.6] | -7.2 [-12.8 to -1.7]
  Day 5: number analyzed (Participants) | 365 | 342
  Day 5 | -4.0 [-11.9 to 3.9] | -8.5 [-13.1 to -4.0]
  Day 8: number analyzed (Participants) | 204 | 193
  Day 8 | -10.8 [-19.8 to -1.8] | -12.0 [-27.6 to 3.6]
  Day 11: number analyzed (Participants) | 126 | 115
  Day 11 | -12.1 [-19.4 to -4.9] | -16.4 [-23.0 to -9.8]
  Day 15: number analyzed (Participants) | 201 | 181
  Day 15 | -13.4 [-19.9 to -6.8] | -15.4 [-20.8 to -10.0]
  Day 29: number analyzed (Participants) | 219 | 191
  Day 29 | -18.6 [-23.8 to -13.4] | 9.9 [-53.3 to 73.2]

4. Secondary Outcome: Change From Baseline in C-reactive Protein (CRP)
Description: Blood to evaluate CRP was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge.
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: The mITT population includes all participants by their randomized treatment assignment and baseline ordinal score. For missing data, if results were available for visits before or after that visit, the average of the two nearest visits was imputed. If a participant died or was lost to follow-up, their last available observation was carried forward. If baseline was missing, the earliest post-treatment dose was used. Participants from sites reporting high sensitivity CRP were excluded.
Measure: Mean (95% Confidence Interval); unit: milligrams/liter (mg/L)
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Dexamethasone
Number analyzed (Participants) | 437 | 415
milligrams/liter (mg/L)
  Day 3 | -41.1 [-46.6 to -35.5] | -61.0 [-66.9 to -55.2]
  Day 5 | -39.4 [-46.0 to -32.8] | -73.6 [-80.1 to -67.0]
  Day 8 | -53.0 [-60.3 to -45.7] | -79.0 [-86.1 to -72.0]
  Day 11 | -61.6 [-69.2 to -54.1] | -81.6 [-88.9 to -74.3]
  Day 15 | -73.2 [-80.8 to -65.7] | -81.1 [-88.7 to -73.4]
  Day 29 | -78.6 [-86.2 to -70.9] | -84.1 [-91.8 to -76.4]

5. Secondary Outcome: Change From Baseline in Creatinine
Description: Blood to evaluate serum creatinine was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge.
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Dexamethasone
Number analyzed (Participants) | 484 | 461
mg/dL
  Day 3 | -0.207 [-0.521 to 0.108] | -0.081 [-0.102 to -0.059]
  Day 5: number analyzed (Participants) | 368 | 346
  Day 5 | -0.287 [-0.701 to 0.127] | -0.122 [-0.147 to -0.097]
  Day 8: number analyzed (Participants) | 206 | 194
  Day 8 | -0.434 [-1.175 to 0.308] | -0.096 [-0.132 to -0.060]
  Day 11: number analyzed (Participants) | 128 | 115
  Day 11 | 0.007 [-0.121 to 0.135] | -0.102 [-0.165 to -0.039]
  Day 15: number analyzed (Participants) | 203 | 185
  Day 15 | -0.011 [-0.101 to 0.080] | -0.024 [-0.086 to 0.039]
  Day 29: number analyzed (Participants) | 222 | 192
  Day 29 | -0.064 [-0.100 to -0.029] | -0.029 [-0.090 to 0.031]

6. Secondary Outcome: Change From Baseline in D-dimer Concentration
Description: Blood to evaluate d-dimer concentration was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge.
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: The mITT population includes all participants by their randomized treatment assignment and baseline ordinal score. For any missing data, if results were available for visits before or after that visit, the average of the two nearest visits was imputed for all missing visits between them. If a participant died or was lost to follow-up, their last available observation was carried forward. If baseline was missing, another pre-treatment dose was used, or the earliest post-treatment dose was used.
Measure: Mean (95% Confidence Interval); unit: mg/L fibrinogen-equivalent units (FEU)
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Dexamethasone
Number analyzed (Participants) | 490 | 467
mg/L fibrinogen-equivalent units (FEU)
  Day 3 | 0.8 [0.3 to 1.3] | 0.2 [-0.1 to 0.6]
  Day 5 | 0.7 [0.3 to 1.1] | 0.7 [0.2 to 1.2]
  Day 8 | 0.7 [0.2 to 1.2] | 0.9 [0.3 to 1.5]
  Day 11 | 0.7 [0.0 to 1.3] | 0.5 [0.0 to 0.9]
  Day 15 | 0.1 [-0.2 to 0.3] | 0.3 [-0.1 to 0.7]
  Day 29 | 0.1 [-0.2 to 0.3] | 0.2 [-0.2 to 0.6]

7. Secondary Outcome: Change From Baseline in Glucose
Description: Blood to evaluate glucose was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge.
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Dexamethasone
Number analyzed (Participants) | 484 | 461
mg/dL
  Day 3 | -46.9 [-53.0 to -40.8] | 3.8 [-2.4 to 10.0]
  Day 5: number analyzed (Participants) | 368 | 346
  Day 5 | -43.2 [-50.9 to -35.5] | -6.7 [-14.9 to 1.5]
  Day 8: number analyzed (Participants) | 206 | 194
  Day 8 | -35.0 [-45.5 to -24.4] | -9.6 [-22.0 to 2.8]
  Day 11: number analyzed (Participants) | 128 | 115
  Day 11 | -28.1 [-43.2 to -13.0] | -15.0 [-30.6 to 0.6]
  Day 15: number analyzed (Participants) | 203 | 185
  Day 15 | -26.0 [-35.3 to -16.6] | -20.2 [-31.3 to -9.1]
  Day 29: number analyzed (Participants) | 222 | 192
  Day 29 | -28.9 [-38.8 to -19.0] | -25.4 [-36.1 to -14.8]

8. Secondary Outcome: Change From Baseline in Hemoglobin
Description: Blood to evaluate hemoglobin was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge.
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: grams/deciliter (g/dL)
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Dexamethasone
Number analyzed (Participants) | 481 | 458
grams/deciliter (g/dL)
  Day 3 | -0.51 [-0.59 to -0.43] | -0.25 [-0.35 to -0.15]
  Day 5: number analyzed (Participants) | 368 | 342
  Day 5 | -0.64 [-0.80 to -0.47] | -0.13 [-0.25 to 0.00]
  Day 8: number analyzed (Participants) | 206 | 194
  Day 8 | -1.08 [-1.28 to -0.88] | -0.15 [-0.37 to 0.07]
  Day 11: number analyzed (Participants) | 130 | 116
  Day 11 | -1.44 [-1.75 to -1.13] | -0.76 [-1.03 to -0.48]
  Day 15: number analyzed (Participants) | 203 | 182
  Day 15 | -0.97 [-1.23 to -0.71] | -0.91 [-1.13 to -0.69]
  Day 29: number analyzed (Participants) | 221 | 186
  Day 29 | -0.51 [-0.75 to -0.28] | -0.66 [-0.93 to -0.39]

9. Secondary Outcome: Change From Baseline in Platelets
Description: Blood to evaluate platelets was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge.
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: 10^9 cells/liter
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Dexamethasone
Number analyzed (Participants) | 479 | 456
10^9 cells/liter
  Day 3 | 53.1 [48.6 to 57.5] | 70.4 [65.6 to 75.1]
  Day 5: number analyzed (Participants) | 366 | 341
  Day 5 | 107.4 [98.8 to 116.0] | 117.6 [108.9 to 126.4]
  Day 8: number analyzed (Participants) | 205 | 193
  Day 8 | 178.9 [161.4 to 196.3] | 140.4 [125.7 to 155.1]
  Day 11: number analyzed (Participants) | 129 | 115
  Day 11 | 193.9 [166.5 to 221.3] | 105.0 [86.7 to 123.4]
  Day 15: number analyzed (Participants) | 203 | 183
  Day 15 | 139.6 [119.0 to 160.3] | 45.3 [29.4 to 61.1]
  Day 29: number analyzed (Participants) | 221 | 186
  Day 29 | 35.3 [22.8 to 47.8] | 69.4 [56.1 to 82.7]

10. Secondary Outcome: Change From Baseline in Prothrombin International Normalized Ratio (INR)
Description: Blood to evaluate INR was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge.
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Dexamethasone
Number analyzed (Participants) | 445 | 412
ratio
  Day 3 | 0.06 [0.04 to 0.09] | -0.01 [-0.08 to 0.06]
  Day 5: number analyzed (Participants) | 326 | 299
  Day 5 | 0.11 [0.09 to 0.13] | -0.03 [-0.13 to 0.07]
  Day 8: number analyzed (Participants) | 183 | 168
  Day 8 | 0.11 [0.08 to 0.14] | -0.08 [-0.25 to 0.09]
  Day 11: number analyzed (Participants) | 112 | 99
  Day 11 | 0.09 [0.03 to 0.14] | -0.14 [-0.42 to 0.14]
  Day 15: number analyzed (Participants) | 180 | 153
  Day 15 | 0.00 [-0.03 to 0.03] | -0.04 [-0.08 to 0.00]
  Day 29: number analyzed (Participants) | 209 | 173
  Day 29 | -0.06 [-0.09 to -0.04] | -0.05 [-0.08 to -0.03]

11. Secondary Outcome: Change From Baseline in Total Bilirubin
Description: Blood to evaluate total bilirubin was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge.
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Dexamethasone
Number analyzed (Participants) | 482 | 458
mg/dL
  Day 3 | 0.00 [-0.02 to 0.02] | -0.09 [-0.11 to -0.07]
  Day 5: number analyzed (Participants) | 365 | 342
  Day 5 | 0.06 [0.03 to 0.08] | -0.03 [-0.06 to 0.01]
  Day 8: number analyzed (Participants) | 204 | 193
  Day 8 | 0.03 [-0.01 to 0.06] | 0.03 [-0.01 to 0.07]
  Day 11: number analyzed (Participants) | 126 | 115
  Day 11 | 0.04 [-0.03 to 0.11] | 0.05 [-0.01 to 0.11]
  Day 15: number analyzed (Participants) | 202 | 182
  Day 15 | -0.01 [-0.06 to 0.04] | 0.03 [-0.02 to 0.08]
  Day 29: number analyzed (Participants) | 219 | 191
  Day 29 | -0.02 [-0.05 to 0.02] | -0.05 [-0.10 to -0.01]

12. Secondary Outcome: Change From Baseline in White Blood Cell Count (WBC)
Description: Blood to evaluate WBC was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge.
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: 10^9 cells/liter
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Dexamethasone
Number analyzed (Participants) | 481 | 458
10^9 cells/liter
  Day 3 | 0.433 [0.196 to 0.670] | 1.292 [1.054 to 1.529]
  Day 5: number analyzed (Participants) | 368 | 342
  Day 5 | 1.358 [1.006 to 1.709] | 2.072 [1.712 to 2.432]
  Day 8: number analyzed (Participants) | 206 | 192
  Day 8 | 2.629 [1.946 to 3.311] | 4.048 [3.415 to 4.681]
  Day 11: number analyzed (Participants) | 130 | 116
  Day 11 | 4.153 [3.098 to 5.209] | 5.179 [4.177 to 6.182]
  Day 15: number analyzed (Participants) | 203 | 183
  Day 15 | 1.638 [0.965 to 2.310] | 2.386 [1.697 to 3.074]
  Day 29: number analyzed (Participants) | 221 | 186
  Day 29 | 0.688 [0.103 to 1.273] | 0.116 [-0.468 to 0.699]

13. Secondary Outcome: Change From Baseline in Neutrophils
Description: Blood to evaluate neutrophils was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge.
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: 10^9 cells/liter
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Dexamethasone
Number analyzed (Participants) | 477 | 451
10^9 cells/liter
  Day 3 | -0.500 [-0.721 to -0.280] | 0.974 [0.749 to 1.200]
  Day 5: number analyzed (Participants) | 364 | 340
  Day 5 | 0.356 [0.007 to 0.704] | 1.407 [1.076 to 1.738]
  Day 8: number analyzed (Participants) | 205 | 192
  Day 8 | 1.421 [0.763 to 2.080] | 3.227 [2.621 to 3.833]
  Day 11: number analyzed (Participants) | 130 | 113
  Day 11 | 2.937 [1.935 to 3.940] | 4.135 [3.177 to 5.093]
  Day 15: number analyzed (Participants) | 201 | 180
  Day 15 | 0.416 [-0.216 to 1.047] | 1.229 [0.560 to 1.898]
  Day 29: number analyzed (Participants) | 221 | 187
  Day 29 | -0.659 [-1.227 to -0.092] | -1.239 [-1.801 to -0.677]

14. Secondary Outcome: Change From Baseline in Lymphocytes
Description: Blood to evaluate lymphocytes was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge.
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: 10^9 cells/liter
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Dexamethasone
Number analyzed (Participants) | 477 | 451
10^9 cells/liter
  Day 3 | 0.766 [0.678 to 0.854] | 0.142 [0.100 to 0.183]
  Day 5: number analyzed (Participants) | 364 | 340
  Day 5 | 0.627 [0.559 to 0.696] | 0.356 [0.293 to 0.420]
  Day 8: number analyzed (Participants) | 205 | 192
  Day 8 | 0.614 [0.517 to 0.712] | 0.317 [0.231 to 0.403]
  Day 11: number analyzed (Participants) | 130 | 113
  Day 11 | 0.594 [0.462 to 0.727] | 0.372 [0.275 to 0.470]
  Day 15: number analyzed (Participants) | 201 | 180
  Day 15 | 0.693 [0.599 to 0.788] | 0.621 [0.536 to 0.706]
  Day 29: number analyzed (Participants) | 221 | 187
  Day 29 | 0.842 [0.650 to 1.033] | 0.996 [0.900 to 1.092]

15. Secondary Outcome: Change From Baseline in Monocytes
Description: Blood to evaluate monocytes was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge.
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: 10^9 cells/liter
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Dexamethasone
Number analyzed (Participants) | 477 | 450
10^9 cells/liter
  Day 3 | 0.114 [0.090 to 0.138] | 0.120 [0.096 to 0.143]
  Day 5: number analyzed (Participants) | 363 | 340
  Day 5 | 0.164 [0.133 to 0.195] | 0.180 [0.148 to 0.213]
  Day 8: number analyzed (Participants) | 205 | 192
  Day 8 | 0.257 [0.208 to 0.306] | 0.221 [0.174 to 0.268]
  Day 11: number analyzed (Participants) | 130 | 113
  Day 11 | 0.367 [0.283 to 0.452] | 0.306 [0.228 to 0.384]
  Day 15: number analyzed (Participants) | 201 | 179
  Day 15 | 0.295 [0.246 to 0.344] | 0.286 [0.232 to 0.340]
  Day 29: number analyzed (Participants) | 221 | 187
  Day 29 | 0.171 [0.133 to 0.209] | 0.159 [0.121 to 0.198]

16. Secondary Outcome: Change From Baseline in Basophils
Description: Blood to evaluate basophils was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge.
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: 10^9 cells/liter
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Dexamethasone
Number analyzed (Participants) | 471 | 446
10^9 cells/liter
  Day 3 | 0.008 [0.005 to 0.011] | 0.000 [-0.003 to 0.002]
  Day 5: number analyzed (Participants) | 357 | 339
  Day 5 | 0.016 [0.011 to 0.020] | 0.004 [0.001 to 0.007]
  Day 8: number analyzed (Participants) | 203 | 192
  Day 8 | 0.015 [0.011 to 0.020] | 0.006 [0.002 to 0.009]
  Day 11: number analyzed (Participants) | 129 | 113
  Day 11 | 0.021 [0.014 to 0.027] | 0.006 [0.000 to 0.012]
  Day 15: number analyzed (Participants) | 199 | 179
  Day 15 | 0.035 [0.029 to 0.041] | 0.030 [0.021 to 0.038]
  Day 29: number analyzed (Participants) | 220 | 187
  Day 29 | 0.043 [0.035 to 0.051] | 0.046 [0.033 to 0.060]

17. Secondary Outcome: Change From Baseline in Eosinophils
Description: Blood to evaluate eosinophils was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge.
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: 10^9 cells/liter
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Dexamethasone
Number analyzed (Participants) | 472 | 446
10^9 cells/liter
  Day 3 | 0.034 [0.029 to 0.040] | -0.006 [-0.009 to -0.002]
  Day 5: number analyzed (Participants) | 357 | 339
  Day 5 | 0.104 [0.092 to 0.116] | 0.006 [0.002 to 0.010]
  Day 8: number analyzed (Participants) | 203 | 192
  Day 8 | 0.115 [0.100 to 0.131] | 0.027 [0.016 to 0.038]
  Day 11: number analyzed (Participants) | 129 | 113
  Day 11 | 0.116 [0.089 to 0.143] | 0.034 [0.020 to 0.049]
  Day 15: number analyzed (Participants) | 199 | 179
  Day 15 | 0.124 [0.108 to 0.141] | 0.119 [0.102 to 0.136]
  Day 29: number analyzed (Participants) | 220 | 187
  Day 29 | 0.208 [0.179 to 0.238] | 0.211 [0.169 to 0.253]

18. Secondary Outcome: Percentage of Participants Reporting Grade 3 and 4 Clinical and/or Laboratory Adverse Events (AEs)
Description: Grade 3 AEs are defined as events that interrupt usual activities of daily living, or significantly affects clinical status, or may require intensive therapeutic intervention. Severe events are usually incapacitating. Grade 4 AEs are defined as events that are potentially life threatening.
Time Frame: Day 1 through Day 29
Population: The safety population includes all participants with available data post baseline, analyzed as treated.
Measure: Number; unit: percentage of participants
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Dexamethasone
Number analyzed (Participants) | 503 | 482
percentage of participants | 28.4 | 36.1
Statistical Analysis 1: Comparison: Remdesivir Plus Baricitinib vs Remdesivir Plus Dexamethasone; Test type: Superiority; Risk Difference (RD) = 7.7, 95% CI 2-sided [1.8 to 13.4]

19. Secondary Outcome: Percentage of Participants Reporting Serious Adverse Events (SAEs)
Description: An SAE is defined as an AE or suspected adverse reaction is considered serious if, in the view of either the investigator or the sponsor, it results in death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or a congenital anomaly/birth defect.
Time Frame: Day 1 through Day 29
Population: The safety population includes all participants with available data post baseline, analyzed as treated.
Measure: Number; unit: percentage of participants
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Dexamethasone
Number analyzed (Participants) | 503 | 482
percentage of participants | 18.9 | 19.5
Statistical Analysis 1: Comparison: Remdesivir Plus Baricitinib vs Remdesivir Plus Dexamethasone; Test type: Superiority; Risk Difference (RD) = 0.6, 95% CI 2-sided [-4.3 to 5.5]

20. Secondary Outcome: Days of Invasive Mechanical Ventilation / Extracorporeal Membrane Oxygenation (ECMO)
Description: Duration of invasive ventilation/ECMO was measured in days among participants who required invasive ventilation, determined two ways. The first includes imputations for participants who died. The second method is restricted to participants who did not die.
Time Frame: Day 1 through Day 29
Population: The analysis population is restricted to randomized participants who were on invasive ventilation.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Dexamethasone
Number analyzed (Participants) | 55 | 47
Days
  Including imputations for participants who died | 27 [14 to 28] | 28 [18 to 28]
  Among participants who did not die: number analyzed (Participants) | 37 | 24
  Among participants who did not die | 14 [8 to 23] | 15 [10 to 20]

21. Secondary Outcome: Days of Non-invasive Ventilation/High Flow Oxygen
Description: Duration of new non-invasive ventilation or high flow oxygen use was measured in days among participants who were not on non-invasive ventilation or high-flow oxygen use at baseline, determined two ways. The first includes imputations for participants who died. The second method is restricted to participants who did not die.
Time Frame: Day 1 through Day 29
Population: The analysis population is restricted to randomized participants who were not on noninvasive ventilation or high-flow oxygen at baseline but who subsequently required non-invasive or high-flow oxygen.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Dexamethasone
Number analyzed (Participants) | 69 | 88
Days
  Including imputations for participants who died | 5 [3 to 9] | 8 [4 to 28]
  Among participants who did not die: number analyzed (Participants) | 61 | 69
  Among participants who did not die | 4 [2 to 7] | 6 [4 to 10]

22. Secondary Outcome: Duration of Supplemental Oxygen Use
Description: Duration of supplemental oxygen use was measured in days among participants who were on oxygen at baseline, calculated in two ways. The first includes imputations for participants who died. The second method is restricted to participants who did not die.
Time Frame: Day 1 through Day 29
Population: The analysis population is restricted to randomized participants who were on oxygen at baseline.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Dexamethasone
Number analyzed (Participants) | 515 | 494
Days
  Including imputations for participants who died | 10 [4 to 28] | 10.5 [4 to 28]
  Among participants who did not die: number analyzed (Participants) | 487 | 460
  Among participants who did not die | 9 [4 to 28] | 8 [4 to 28]

23. Secondary Outcome: Desirability of Outcome Ranking (DOOR) at Day 15
Description: Desirability of Outcome Ranking (DOOR) based on ordinal scale: 1) Recovered (category 1, 2 or 3 on ordinal scale); 2) Improved (> / = 1 category improvement of ordinal scale compared with baseline) & no serious adverse event (SAE); 3) Improved (> / = 1 category improvement of the ordinal scale compared with baseline) & SAE (related or unrelated); 4) No change in ordinal scale from baseline & no SAE; 5) No change in ordinal scale from baseline & SAE (related or unrelated); 6) Worsening (> / = 1 category worse in ordinal scale from baseline); 7) Death.
Time Frame: Day 1 through Day 15
Population: The modified intention-to-treat (mITT) population includes all participants who were randomized, classified by their randomized treatment assignment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Dexamethasone
Number analyzed (Participants) | 515 | 494
percentage of participants
  1 - Recovered (Category 1, 2 or 3 Clinical Status) | 76 [71.8 to 79.2] | 77 [73.0 to 80.4]
  2 - Improved (=1 category improvement in Clinical Status compared with baseline) & no SAE | 3 [1.5 to 4.3] | 1 [0.4 to 2.3]
  3 - Improved (=1 category improvement compared with baseline) & SAE (related or unrelated) | 1 [0.5 to 2.5] | 2 [1.0 to 3.4]
  4 - No change in Clinical Status from baseline & no SAE | 7 [5.3 to 9.7] | 6 [4.3 to 8.5]
  5 - No change in Clinical Status from baseline & SAE (related or unrelated) | 3 [2.2 to 5.5] | 2 [1.1 to 3.7]
  6 - Worsening (=1 category worse in Clinical Status compared with baseline) | 7 [4.9 to 9.3] | 10 [7.2 to 12.4]
  7 - Death | 3 [1.9 to 5.0] | 3 [1.5 to 4.4]

24. Secondary Outcome: Desirability of Outcome Ranking (DOOR) at Day 29
Description: as for outcome 23
Time Frame: Day 1 through Day 29
Population: as for outcome 23
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Dexamethasone
Number analyzed (Participants) | 515 | 494
percentage of participants
  1 - Recovered (Category 1, 2 or 3 Clinical Status) | 85 [81.5 to 87.7] | 84 [80.5 to 87.0]
  2 - Improved (=1 category improvement in Clinical Status compared with baseline) & no SAE | 0.002 [0.0 to 1.1] | 0.002 [0.0 to 1.1]
  3 - Improved (=1 category improvement compared with baseline) & SAE (related or unrelated) | 1 [0.7 to 2.8] | 1 [0.4 to 2.3]
  4 - No change in Clinical Status from baseline & no SAE | 3 [2.1 to 5.2] | 3 [2.0 to 5.2]
  5 - No change in Clinical Status from baseline & SAE (related or unrelated) | 1 [0.7 to 2.8] | 1 [0.2 to 1.8]
  6 - Worsening (=1 category worse in Clinical Status compared with baseline) | 3 [2.2 to 5.5] | 4 [2.6 to 6.2]
  7 - Death | 5 [3.8 to 7.7] | 7 [5.0 to 9.5]

25. Secondary Outcome: Duration of Hospitalization
Description: Duration of hospitalization was determined two ways. The first includes imputations for participants who died. The second method is restricted to participants who did not die.
Time Frame: Day 1 through Day 29
Population: The modified intent-to-treat (ITT) population includes all participants who were randomized, classified by their randomized treatment assignment.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Dexamethasone
Number analyzed (Participants) | 515 | 494
Days
  Including imputations for participants who died | 7 [4 to 12] | 6 [4 to 11]
  Among participants who did not die: number analyzed (Participants) | 487 | 460
  Among participants who did not die | 6 [4 to 10] | 6 [4 to 9]

26. Secondary Outcome: Number of Participants With Discontinuation or Temporary Suspension of Study Product Administration
Description: Discontinuation or temporary suspension of study product administration, including participants who died or were discharged, was evaluated for each study product/placebo.
Time Frame: Day 1 through Day 10
Population: The mITT population includes all participants who were randomized, classified by their randomized treatment assignment.
Measure: Count of Participants; unit: Participants
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Dexamethasone
Number analyzed (Participants) | 516 | 494
Participants
  Remdesivir | 460 | 444
  Baricitinib/Placebo | 486 | 452
  Dexamethasone/placebo | 410 | 387

27. Secondary Outcome: 14-day Participant Mortality
Description: The mortality rate was determined as the proportion of participants who died by study Day 15. The proportions reported are Kaplan-Meier estimates.
Time Frame: Day 1 through Day 15
Population: The mITT population includes all participants who were randomized, classified by their randomized treatment assignment.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Dexamethasone
Number analyzed (Participants) | 516 | 494
Proportion of participants | 0.03 [0.02 to 0.05] | 0.02 [0.01 to 0.04]

28. Secondary Outcome: 28-day Participant Mortality
Description: The mortality rate was determined as the proportion of participants who died by study Day 29. The proportions reported are Kaplan-Meier estimates.
Time Frame: Day 1 through Day 29
Population: The mITT population includes all participants who were randomized, classified by their randomized treatment assignment.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Dexamethasone
Number analyzed (Participants) | 516 | 494
Proportion of participants | 0.05 [0.04 to 0.08] | 0.06 [0.05 to 0.09]

29. Secondary Outcome: Percentage of Participants at Each Clinical Status Using Ordinal Scale at Day 1
Description: The ordinal scale is an assessment of the clinical status at the first assessment of a given study day. The scale is as follows: 8) Death; 7) Hospitalized, on invasive mechanical ventilation or ECMO; 6) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 5) Hospitalized, requiring supplemental oxygen; 4) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 3) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 2) Not hospitalized, but has new or increased limitation on activities and/or new or increased requirement for home oxygen over baseline, pre-COVID-19 status; 1) Not hospitalized, participant is back to their baseline, pre-COVID-19 status, that is, no new or increased limitations on activities and no new or increased oxygen use.
Time Frame: Day 1
Population: The mITT population includes all participants who were randomized, classified by their randomized treatment assignment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Dexamethasone
Number analyzed (Participants) | 515 | 494
percentage of participants
  8) Death | 0.2 [0.0 to 1.1] | 0.0 [0.0 to 0.8]
  7) Hospitalized, on invasive mechanical ventilation or ECMO | 0.0 [0.0 to 0.7] | 0.0 [0.0 to 0.8]
  6) Hospitalized, on non-invasive ventilation or high flow oxygen devices | 16.1 [13.2 to 19.5] | 14.2 [11.4 to 17.5]
  5) Hospitalized, requiring supplemental oxygen | 83.7 [80.3 to 86.6] | 85.8 [82.5 to 88.6]
  4) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care | 0.0 [0.0 to 0.7] | 0.0 [0.0 to 0.8]
  3) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care | 0.0 [0.0 to 0.7] | 0.0 [0.0 to 0.8]
  2) Not hospitalized, but has new or increased limitation on activities and/or need for oxygen | 0.0 [0.0 to 0.7] | 0.0 [0.0 to 0.8]
  1) Not hospitalized, no limitations on activities | 0.0 [0.0 to 0.7] | 0.0 [0.0 to 0.8]

30. Secondary Outcome: Percentage of Participants at Each Clinical Status Using Ordinal Scale at Day 3
Description: as for outcome 29
Time Frame: Day 3
Population: as for outcome 23
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Dexamethasone
Number analyzed (Participants) | 515 | 494
percentage of participants
  8) Death | 0.4 [0.1 to 1.4] | 0.4 [0.1 to 1.5]
  7) Hospitalized, on invasive mechanical ventilation or ECMO | 3.1 [1.9 to 5.0] | 1.0 [0.4 to 2.3]
  6) Hospitalized, on non-invasive ventilation or high flow oxygen devices | 22.1 [18.8 to 25.9] | 21.5 [18.1 to 25.3]
  5) Hospitalized, requiring supplemental oxygen | 71.7 [67.6 to 75.4] | 73.5 [69.4 to 77.2]
  4) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care | 2.7 [1.6 to 4.5] | 3.2 [2.0 to 5.2]
  3) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care | 0.0 [0.0 to 0.7] | 0.0 [0.0 to 0.8]
  2) Not hospitalized, but has new or increased limitation on activities and/or need for oxygen | 0.0 [0.0 to 0.7] | 0.4 [0.1 to 1.5]
  1) Not hospitalized, no limitations on activities | 0.0 [0.0 to 0.7] | 0.0 [0.0 to 0.8]

31. Secondary Outcome: Percentage of Participants at Each Clinical Status Using Ordinal Scale at Day 5
Description: as for outcome 29
Time Frame: Day 5
Population: as for outcome 23
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Dexamethasone
Number analyzed (Participants) | 515 | 494
percentage of participants
  8) Death | 0.6 [0.2 to 1.7] | 0.4 [0.1 to 1.5]
  7) Hospitalized, on invasive mechanical ventilation or ECMO | 5.2 [3.6 to 7.5] | 3.4 [2.2 to 5.4]
  6) Hospitalized, on non-invasive ventilation or high flow oxygen devices | 19.4 [16.2 to 23.1] | 20.9 [17.5 to 24.7]
  5) Hospitalized, requiring supplemental oxygen | 53.4 [49.1 to 57.7] | 49.2 [44.8 to 53.6]
  4) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care | 9.5 [7.3 to 12.4] | 11.9 [9.4 to 15.1]
  3) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care | 1.2 [0.5 to 2.5] | 0.6 [0.2 to 1.8]
  2) Not hospitalized, but has new or increased limitation on activities and/or need for oxygen | 10.7 [8.3 to 13.6] | 13.2 [10.5 to 16.4]
  1) Not hospitalized, no limitations on activities | 0.0 [0.0 to 0.7] | 0.4 [0.1 to 1.5]

32. Secondary Outcome: Percentage of Participants at Each Clinical Status Using Ordinal Scale at Day 8
Description: as for outcome 29
Time Frame: Day 8
Population: as for outcome 23
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Dexamethasone
Number analyzed (Participants) | 515 | 494
percentage of participants
  8) Death | 1.2 [0.5 to 2.5] | 0.8 [0.3 to 2.1]
  7) Hospitalized, on invasive mechanical ventilation or ECMO | 7.4 [5.4 to 10.0] | 6.1 [4.3 to 8.5]
  6) Hospitalized, on non-invasive ventilation or high flow oxygen devices | 12.2 [9.7 to 15.3] | 14.6 [11.7 to 18.0]
  5) Hospitalized, requiring supplemental oxygen | 24.9 [21.3 to 28.8] | 24.5 [20.9 to 28.5]
  4) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care | 6.4 [4.6 to 8.9] | 5.7 [4.0 to 8.1]
  3) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care | 1.4 [0.7 to 2.8] | 1.4 [0.7 to 2.9]
  2) Not hospitalized, but has new or increased limitation on activities and/or need for oxygen | 46.4 [42.1 to 50.7] | 47.0 [42.6 to 51.4]
  1) Not hospitalized, no limitations on activities | 0.2 [0.0 to 1.1] | 0.0 [0.0 to 0.8]

33. Secondary Outcome: Percentage of Participants at Each Clinical Status Using Ordinal Scale at Day 11
Description: as for outcome 29
Time Frame: Day 11
Population: as for outcome 23
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Dexamethasone
Number analyzed (Participants) | 515 | 494
percentage of participants
  8) Death | 2.1 [1.2 to 3.8] | 1.2 [0.6 to 2.6]
  7) Hospitalized, on invasive mechanical ventilation or ECMO | 7.8 [5.8 to 10.4] | 6.9 [5.0 to 9.5]
  6) Hospitalized, on non-invasive ventilation or high flow oxygen devices | 6.6 [4.8 to 9.1] | 9.1 [6.9 to 12.0]
  5) Hospitalized, requiring supplemental oxygen | 14.4 [11.6 to 17.7] | 11.1 [8.7 to 14.2]
  4) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care | 2.7 [1.6 to 4.5] | 3.2 [2.0 to 5.2]
  3) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care | 1.4 [0.7 to 2.8] | 0.4 [0.1 to 1.5]
  2) Not hospitalized, but has new or increased limitation on activities and/or need for oxygen | 63.5 [59.3 to 67.5] | 66.4 [62.1 to 70.4]
  1) Not hospitalized, no limitations on activities | 1.6 [0.8 to 3.0] | 1.6 [0.8 to 3.2]

34. Secondary Outcome: Percentage of Participants at Each Clinical Status Using Ordinal Scale at Day 15
Description: as for outcome 29
Time Frame: Day 15
Population: as for outcome 23
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Dexamethasone
Number analyzed (Participants) | 515 | 494
percentage of participants
  8) Death | 3.1 [1.9 to 5.0] | 2.6 [1.5 to 4.4]
  7) Hospitalized, on invasive mechanical ventilation or ECMO | 6.2 [4.4 to 8.6] | 6.1 [4.3 to 8.5]
  6) Hospitalized, on non-invasive ventilation or high flow oxygen devices | 3.7 [2.4 to 5.7] | 5.3 [3.6 to 7.6]
  5) Hospitalized, requiring supplemental oxygen | 9.3 [7.1 to 12.1] | 7.9 [5.8 to 10.6]
  4) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care | 1.9 [1.1 to 3.5] | 1.2 [0.6 to 2.6]
  3) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care | 1.0 [0.4 to 2.3] | 0.4 [0.1 to 1.5]
  2) Not hospitalized, but has new or increased limitation on activities and/or need for oxygen | 51.5 [47.1 to 55.7] | 53.6 [49.2 to 58.0]
  1) Not hospitalized, no limitations on activities | 23.3 [19.9 to 27.1] | 22.9 [19.4 to 26.8]

35. Secondary Outcome: Percentage of Participants at Each Clinical Status Using Ordinal Scale at Day 22
Description: as for outcome 29
Time Frame: Day 22
Population: as for outcome 23
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Dexamethasone
Number analyzed (Participants) | 515 | 494
percentage of participants
  8) Death | 4.9 [3.3 to 7.1] | 4.9 [3.3 to 7.1]
  7) Hospitalized, on invasive mechanical ventilation or ECMO | 4.3 [2.8 to 6.4] | 4.9 [3.3 to 7.1]
  6) Hospitalized, on non-invasive ventilation or high flow oxygen devices | 2.1 [1.2 to 3.8] | 2.8 [1.7 to 4.7]
  5) Hospitalized, requiring supplemental oxygen | 5.4 [3.8 to 7.7] | 5.5 [3.8 to 7.8]
  4) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care | 0.8 [0.3 to 2.0] | 0.2 [0.0 to 1.1]
  3) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care | 0.0 [0.0 to 0.7] | 0.2 [0.0 to 1.1]
  2) Not hospitalized, but has new or increased limitation on activities and/or need for oxygen | 48.0 [43.7 to 52.3] | 48.0 [43.6 to 52.4]
  1) Not hospitalized, no limitations on activities | 34.6 [30.6 to 38.8] | 33.6 [29.6 to 37.9]

36. Secondary Outcome: Percentage of Participants at Each Clinical Status Using Ordinal Scale at Day 29
Description: as for outcome 29
Time Frame: Day 29
Population: as for outcome 23
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Dexamethasone
Number analyzed (Participants) | 515 | 494
percentage of participants
  8) Death | 5.4 [3.8 to 7.7] | 6.9 [5.0 to 9.5]
  7) Hospitalized, on invasive mechanical ventilation or ECMO | 2.7 [1.6 to 4.5] | 2.6 [1.5 to 4.4]
  6) Hospitalized, on non-invasive ventilation or high flow oxygen devices | 2.3 [1.3 to 4.0] | 2.6 [1.5 to 4.4]
  5) Hospitalized, requiring supplemental oxygen | 4.1 [2.7 to 6.2] | 3.4 [2.2 to 5.4]
  4) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care | 0.6 [0.2 to 1.7] | 0.4 [0.1 to 1.5]
  3) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care | 0.0 [0.0 to 0.7] | 0.0 [0.0 to 0.8]
  2) Not hospitalized, but has new or increased limitation on activities and/or need for oxygen | 57.3 [53.0 to 61.5] | 52.0 [47.6 to 56.4]
  1) Not hospitalized, no limitations on activities | 27.6 [23.9 to 31.6] | 32.0 [28.0 to 36.2]

37. Secondary Outcome: Percentage of Participants Meeting Criteria for Each of the 8 Ordinal Scale Categories
Description: The ordinal scale categories are defined as: 8) Death; 7) Hospitalized, on invasive mechanical ventilation or ECMO; 6) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 5) Hospitalized, requiring supplemental oxygen; 4) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 3) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 2) Not hospitalized, but has new or increased limitation on activities and/or new or increased requirement for home oxygen over baseline, pre-COVID-19 status; 1) Not hospitalized, patient is back to their baseline, pre-COVID-19 status, that is, no new or increased limitations on activities and no new or increased oxygen use.
Time Frame: Day 15
Population: as for outcome 23
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Dexamethasone
Number analyzed (Participants) | 515 | 494
Percentage of participants
  8) Death | 3 [1.9 to 5.0] | 3 [1. to 4.4]
  7) Hospitalized, on invasive mechanical ventilation or ECMO | 6 [4.4 to 8.6] | 6 [4.3 to 8.5]
  6) Hospitalized, on non-invasive ventilation or high flow oxygen devices | 4 [2.4 to 5.7] | 5 [3.6 to 7.6]
  5) Hospitalized, requiring supplemental oxygen | 9 [7.1 to 12.1] | 8 [5.8 to 10.6]
  4) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care | 2 [1.1 to 3.5] | 1 [0.6 to 2.6]
  3) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care | 1 [0.4 to 2.3] | 0.4 [0.1 to 1.5]
  2) Not hospitalized, but has new or increased limitation on activities and/or new oxygen use | 51 [47.1 to 55.7] | 54 [49.2 to 58.0]
  1) Not hospitalized, no limitations on activities | 23 [19.9 to 27.1] | 23 [19.4 to 26.8]
Statistical Analysis 1: Comparison: Remdesivir Plus Baricitinib vs Remdesivir Plus Dexamethasone; Test type: Superiority; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.80 to 1.27]

38. Secondary Outcome: The Proportion of Participants Not Meeting Criteria for One of the Three Most Severe Ordinal Scale Categories at Any Time.
Description: The three most severe ordinal scale categories are: 8) Death; 7) Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 6) Hospitalized, on non-invasive ventilation or high flow oxygen devices.
Time Frame: Day 1 through Day 29
Population: as for outcome 23
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Dexamethasone
Number analyzed (Participants) | 432 | 424
Proportion of participants | 0.81 [0.77 to 0.85] | 0.78 [0.74 to 0.82]
Statistical Analysis 1: Comparison: Remdesivir Plus Baricitinib vs Remdesivir Plus Dexamethasone; Test type: Superiority; Risk Difference (RD) = -0.03, 95% CI 2-sided [-0.09 to 0.02]

39. Secondary Outcome: Time to an Improvement of One Category From Baseline Using an Ordinal Scale
Description: The ordinal scale is an assessment of the clinical status at the first assessment of a given study day. The scale is as follows: 8) Death; 7) Hospitalized, on invasive mechanical ventilation or ECMO; 6) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 5) Hospitalized, requiring supplemental oxygen; 4) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 3) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 2) Not hospitalized, but has new or increased limitation on activities and/or new or increased requirement for home oxygen over baseline, pre-COVID-19 status; 1) Not hospitalized, patient is back to their baseline, pre-COVID-19 status, that is, no new or increased limitations on activities and no new or increased oxygen use. Time to improvement by at least one category was determined for each participant.
Time Frame: Day 1 through Day 29
Population: as for outcome 23
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Dexamethasone
Number analyzed (Participants) | 515 | 494
Days | 5.0 [4.0 to 5.0] | 4.0 [4.0 to 5.0]
Statistical Analysis 1: Comparison: Remdesivir Plus Baricitinib vs Remdesivir Plus Dexamethasone; Test type: Superiority; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.94 to 1.23]

40. Secondary Outcome: Time to an Improvement of Two Categories From Baseline Using an Ordinal Scale
Description: The ordinal scale is an assessment of the clinical status at the first assessment of a given study day. The scale is as follows: 8) Death; 7) Hospitalized, on invasive mechanical ventilation or ECMO; 6) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 5) Hospitalized, requiring supplemental oxygen; 4) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 3) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 2) Not hospitalized, but has new or increased limitation on activities and/or new or increased requirement for home oxygen over baseline, pre-COVID-19 status; 1) Not hospitalized, patient is back to their baseline, pre-COVID-19 status, that is, no new or increased limitations on activities and no new or increased oxygen use. Time to improvement by at least two categories was determined for each participant.
Time Frame: Day 1 through Day 29
Population: as for outcome 23
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Dexamethasone
Number analyzed (Participants) | 515 | 494
Days | 6.0 [5.0 to 6.0] | 5.0 [5.0 to 6.0]
Statistical Analysis 1: Comparison: Remdesivir Plus Baricitinib vs Remdesivir Plus Dexamethasone; Test type: Superiority; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.94 to 1.23]

41. Secondary Outcome: Time to Recovery
Description: Day of recovery is defined as the first day on which the participant satisfies one of the following three ordinal scale categories: 3) Hospitalized, not requiring supplemental oxygen and no longer requires ongoing medical care; 2) Not hospitalized, but has new or increased limitation on activities and/or new or increased requirement for home oxygen over baseline, pre-COVID-19 status; 1) Not hospitalized, patient is back to their baseline, pre-COVID-19 status, that is, no new or increased limitations on activities and no new or increased oxygen use.
Time Frame: Day 1 through Day 29
Population: as for outcome 23
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Dexamethasone
Number analyzed (Participants) | 515 | 494
Days | 6.0 [4.0 to 10.0] | 5.0 [3.0 to 9.0]
Statistical Analysis 1: Comparison: Remdesivir Plus Baricitinib vs Remdesivir Plus Dexamethasone; Test type: Superiority; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.91 to 1.19]

42. Primary Outcome: The Proportion of Participants Not Meeting Criteria for One of the Following Two Ordinal Scale Categories at Any Time: 8) Death; 7) Hospitalized, on Invasive Mechanical Ventilation or Extracorporeal Membrane Oxygenation (ECMO) by Race
Description: as for outcome 1
Time Frame: Day 1 through Day 29
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Dexamethasone
Number analyzed (Participants) | 515 | 494
Proportion of participants
  Asian: number analyzed (Participants) | 35 | 35
  Asian | 0.76 [0.58 to 0.87] | 0.88 [0.71 to 0.95]
  Black or African American: number analyzed (Participants) | 94 | 94
  Black or African American | 0.91 [0.83 to 0.96] | 0.86 [0.77 to 0.92]
  White: number analyzed (Participants) | 306 | 281
  White | 0.87 [0.82 to 0.90] | 0.88 [0.83 to 0.91]
  Other: number analyzed (Participants) | 80 | 84
  Other | 0.87 [0.78 to 0.93] | 0.89 [0.80 to 0.94]

43. Primary Outcome: The Proportion of Participants Not Meeting Criteria for One of the Following Two Ordinal Scale Categories at Any Time: 8) Death; 7) Hospitalized, on Invasive Mechanical Ventilation or Extracorporeal Membrane Oxygenation (ECMO) by Ethnicity
Description: as for outcome 1
Time Frame: Day 1 through Day 29
Population: The modified intention-to-treat (mITT) population includes all participants who were randomized and for whom ethnicity was reported. mITT participants were classified by their randomized treatment assignment and their baseline ordinal score, which is not necessarily equivalent to the disease severity stratum to which the participant was randomized at enrollment. One participant was excluded from mITT analyses due to a baseline ordinal score of 4.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Dexamethasone
Number analyzed (Participants) | 505 | 477
Proportion of participants
  Not Hispanic or Latino: number analyzed (Participants) | 317 | 318
  Not Hispanic or Latino | 0.87 [0.82 to 0.90] | 0.87 [0.83 to 0.91]
  Hispanic or Latino: number analyzed (Participants) | 188 | 159
  Hispanic or Latino | 0.88 [0.82 to 0.92] | 0.87 [0.81 to 0.92]

44. Primary Outcome: The Proportion of Participants Not Meeting Criteria for One of the Following Two Ordinal Scale Categories at Any Time: 8) Death; 7) Hospitalized, on Invasive Mechanical Ventilation or Extracorporeal Membrane Oxygenation (ECMO) by Sex
Description: as for outcome 1
Time Frame: Day 1 through Day 29
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Dexamethasone
Number analyzed (Participants) | 515 | 494
Proportion of participants
  Male: number analyzed (Participants) | 299 | 290
  Male | 0.86 [0.81 to 0.89] | 0.87 [0.83 to 0.91]
  Female: number analyzed (Participants) | 216 | 204
  Female | 0.89 [0.84 to 0.93] | 0.88 [0.82 to 0.92]

ADVERSE EVENTS:
Time Frame: Serious and Grade 3 and 4 non-serious adverse events were collected for 29 days after the first dose. Laboratory values were systematically assessed at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29. Treatment emergent and fatal AEs are reported.
Description: Given the severity of underlying illness, participants were expected to have many symptoms and abnormalities in vital signs and laboratory values. All Grade 3 and 4 AEs were captured as AEs in this trial.
  Grade 2 or higher, suspected drug-related hypersensitivity reaction or deep vein thrombosis or pulmonary embolism of any grade was reported as an AE in this trial. All cause mortality was calculated for the ITT population, while SAEs and AEs reflect the as treated population.
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Dexamethasone
All-Cause Mortality (participants affected / at risk) | 28/516 | 34/494
Serious Adverse Events (participants affected / at risk) | 95/503 | 94/482
Other Adverse Events (participants affected / at risk) | 16/503 | 34/482
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Remdesivir Plus Baricitinib (N=503) | Remdesivir Plus Dexamethasone (N=482)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Hypercoagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (2) | 2 (2)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Retinal artery occlusion (Eye disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 2 (2) | 7 (7)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Fungal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 8 (8) | 3 (3)
Pneumonia bacterial (Infections and infestations) | 3 (3) | 3 (3)
Pneumonia klebsiella (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 3 (4) | 4 (4)
Septic shock (Infections and infestations) | 6 (6) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 2 (2) | 2 (2)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 3 (3) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Substance use disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 9 (9) | 4 (4)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 16 (16)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 8 (8)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 10 (10)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 52 (52) | 40 (40)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Remdesivir Plus Baricitinib (N=503) | Remdesivir Plus Dexamethasone (N=482)
Lymphocyte count decreased (Investigations) | 16 (17) | 34 (38)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol (2021-01-18): https://cdn.clinicaltrials.gov/large-docs/68/NCT04640168/Prot_001.pdf
  • Statistical Analysis Plan (2021-06-09): https://cdn.clinicaltrials.gov/large-docs/68/NCT04640168/SAP_003.pdf
  • Informed Consent Form (2021-01-22): https://cdn.clinicaltrials.gov/large-docs/68/NCT04640168/ICF_000.pdf